CLINICAL TRIAL: NCT02878330
Title: A Phase 2b Randomized, Double-Blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of MEDI8897, a Monoclonal Antibody With an Extended Half-life Against Respiratory Syncytial Virus, in Healthy Preterm Infants
Brief Title: A Study to Evaluate the Safety and Efficacy of MEDI8897 for the Prevention of Medically Attended RSV LRTI in Healthy Preterm Infants.
Acronym: MEDI8897 Ph2b
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D5290C00003
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus, RSV; Preterm Infants; Lower Respiratory Tract Infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Participants will receive a single intramuscular (IM) dose of placebo matched to MEDI8897 on Day 1 of the study.
  Interventions: Drug: Placebo
- MEDI8897 50 mg (Experimental): Participants will receive a single IM dose of MEDI8897 50 milligrams (mg) on Day 1 of the study.
  Interventions: Drug: MEDI8897

INTERVENTIONS:
Drug: MEDI8897 — A single IM dose of 50 mg on Day 1 of the study.
  Arms: MEDI8897 50 mg
Drug: Placebo — A single IM dose of placebo matched to MEDI8897 on Day 1 of the study.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy, safety, pharmacokinetics (PK), and antidrug antibody (ADA) response for MEDI8897 in healthy preterm infants who are between 29 and 35 weeks gestational age (GA) and entering their first Respiratory Syncytial Virus (RSV) season.

DETAILED DESCRIPTION:
This pivotal Phase 2b study will determine if MEDI8897 will be efficacious in reducing medically attended RSV-confirmed lower respiratory tract infections (LRTI) in healthy preterm infants entering their first RSV season. The population to be enrolled is healthy preterm infants born between 29 weeks 0 days and 34 weeks 6 days GA who would not receive RSV prophylaxis. A total of 1500 infants will be randomized 2:1 to receive either MEDI8897 or placebo. Participants will be followed for 360 days after dosing. Enrollment is planned at approximately 197 sites across the USA, Canada, Europe, and the Southern Hemisphere.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy infants born between 29 weeks 0 days and 34 weeks 6 days GA.
2. Infants who are entering their first full RSV season at the time of screening.

Key Exclusion Criteria:

1. Meets American Academy of Pediatrics (AAP) or other local criteria to receive commercial palivizumab.
2. Any fever (>= 100.4°F [>= 38.0°C], regardless of route) or lower respiratory illness within 7 days prior to randomization.
3. Acute illness (defined as the presence of moderate or severe signs and symptoms) at the time of randomization.
4. Active RSV infection (a child with signs/symptoms of respiratory infection must have negative RSV testing) or known prior history of RSV infection.
5. Receipt of palivizumab or other RSV monoclonal antibody or any RSV vaccine, including maternal RSV vaccination.

Max Age: 365 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1453 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-12-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (142):
- United States (56):
  - Research Site, Birmingham, Alabama
  - Research Site, Anaheim, California
  - Research Site, Downey, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Paramount, California
  - Research Site, San Diego, California
  - Research Site, West Covina, California
  - Research Site, Aurora, Colorado
  - Research Site, Colorado Springs, Colorado
  - Research Site, Hartford, Connecticut
  - Research Site, Gainesville, Florida
  - Research Site, Orlando, Florida
  - Research Site, South Miami, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Oak Lawn, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, South Bend, Indiana
  - Research Site, Woburn, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site, Mineola, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Stony Brook, New York
  - Research Site, Syracuse, New York
  - Research Site, Boone, North Carolina
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Gresham, Oregon
  - Research Site, Erie, Pennsylvania
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Sioux Falls, South Dakota
  - Research Site, Memphis, Tennessee
  - Research Site, Edinburg, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Galveston, Texas
  - Research Site, Longview, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Layton, Utah
  - Research Site, Orem, Utah
  - Research Site, Syracuse, Utah
  - Research Site, Seattle, Washington
  - Research Site, Huntington, West Virginia
  - Research Site, Morgantown, West Virginia
  - Research Site, Madison, Wisconsin
- Argentina (2):
  - Research Site, Bahía Blanca
  - Research Site, Guaymallen Mendoza
- Australia (2):
  - Research Site, Parkville
  - Research Site, Subiaco
- Belgium (2):
  - Research Site, Ghent
  - Research Site, Mons
- Brazil (6):
  - Research Site, Botucatu
  - Research Site, Campinas
  - Research Site, Canoas
  - Research Site, Curitiba
  - Research Site, Juiz de Fora
  - Research Site, Passo Fundo
- Bulgaria (4):
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Rousse
  - Research Site, Sofia
- Research Site, Montreal, Quebec, Canada
- Chile (4):
  - Research Site, Maipú
  - Research Site, Santiago
  - Research Site, Valdivia
  - Research Site, Viña del Mar
- Czechia (2):
  - Research Site, Havlíčkův Brod
  - Research Site, Prague
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Finland (2):
  - Research Site, Tampere
  - Research Site, Turku
- France (6):
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Dijon
  - Research Site, Tours
- Hungary (10):
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Kecskemét
  - Research Site, Miskolc
  - Research Site, Nagykanizsa
  - Research Site, Nyireyghaza
  - Research Site, Sopron
  - Research Site, Szeged
  - Research Site, Szekszárd
  - Research Site, Veszprém
- Italy (4):
  - Research Site, Genova
  - Research Site, Padua
  - Research Site, Torino
  - Research Site, Verona
- Latvia (3):
  - Research Site, Jēkabpils
  - Research Site, Riga
  - Research Site, Valmiera
- Research Site, Kaunas, Lithuania
- New Zealand (3):
  - Research Site, Christchurch
  - Research Site, Otahuhu
  - Research Site, Wellington
- Poland (4):
  - Research Site, Bydgoszcz
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Łęczna
- South Africa (6):
  - Research Site, Cape Town
  - Research Site, Claremont
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, Pietermaritzburg
  - Research Site, Pretoria
- Spain (11):
  - Research Site, Alicante
  - Research Site, Boadilla del Monte
  - Research Site, Córdoba
  - Research Site, Granada
  - Research Site, Lleida
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Sant Cugat del Vallès
  - Research Site, Sant Joan d'Alacant
  - Research Site, Santiago de Compostela
  - Research Site, Valencia
- Research Site, Stockholm, Sweden
- Turkey (Türkiye) (5):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Izmir
  - Research Site, Kocaeli
- United Kingdom (5):
  - Research Site, Brighton
  - Research Site, Bristol
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Southampton

REFERENCES:
- [Derived] Langer S, Holzapfel S, August L, Badura A, Wellmann S, Mack I. Parental knowledge and attitudes to infant immunization in the context of RSV: All about confidence? Vaccine. 2024 Oct 3;42(23):126050. doi: 10.1016/j.vaccine.2024.06.018. Epub 2024 Jun 19. PMID 38902186
- [Derived] Ahani B, Tuffy KM, Aksyuk AA, Wilkins D, Abram ME, Dagan R, Domachowske JB, Guest JD, Ji H, Kushnir A, Leach A, Madhi SA, Mankad VS, Simoes EAF, Sparklin B, Speer SD, Stanley AM, Tabor DE, Hamren UW, Kelly EJ, Villafana T. Molecular and phenotypic characteristics of RSV infections in infants during two nirsevimab randomized clinical trials. Nat Commun. 2023 Jul 19;14(1):4347. doi: 10.1038/s41467-023-40057-8. PMID 37468530
- [Derived] Griffin MP, Yuan Y, Takas T, Domachowske JB, Madhi SA, Manzoni P, Simoes EAF, Esser MT, Khan AA, Dubovsky F, Villafana T, DeVincenzo JP; Nirsevimab Study Group. Single-Dose Nirsevimab for Prevention of RSV in Preterm Infants. N Engl J Med. 2020 Jul 30;383(5):415-425. doi: 10.1056/NEJMoa1913556. PMID 32726528
- See also: D5290C00003_Redacted_protocol-amendment-1_Red16JLU19 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00003&attachmentIdentifier=b9e98653-9f94-46e7-a735-9a742e555af6&fileName=D5290C00003_Redacted_protocol-amendment-1_Red16JLU19.pdf&versionIdentifier=
- See also: D5290C00003_MEDI8897-Combined SAP_PDFAv1.0 — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5290C00003&attachmentIdentifier=f0ccb086-5c35-4e3c-9dde-0fefc3989cd9&fileName=D5290C00003_MEDI8897-Combined_SAP_PDFAv1.0.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 03-Nov-2016 to 06-Dec-2018.
Pre-assignment Details: A total of 1540 participants were screened, out of which 1453 participants were randomized in the study.
Groups:
- Placebo: Participants received a single intramuscular (IM) dose of placebo matched to MEDI8897 on Day 1 of the study.
- MEDI8897 50 mg: Participants received a single IM dose of MEDI8897 50 milligrams (mg) on Day 1 of the study.
Period: Overall Study
Arm/Group | Placebo | MEDI8897 50 mg
Started | 484 | 969
Completed | 455 | 913
Not Completed | 29 | 56
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 11 | 26
Not completed — Withdrawal by Subject | 11 | 21
Not completed — Other | 4 | 7

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were randomized in the study and analyzed according to their randomized treatment group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MEDI8897 50 mg | Total
Number analyzed (Participants) | 484 | 969 | 1453
Age, Continuous [Mean (Standard Deviation); unit: Months] | 3.28 (2.31) | 3.29 (2.22) | 3.29 (2.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 468 | 692
  Male | 260 | 501 | 761
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 225 | 316
  Not Hispanic or Latino | 393 | 743 | 1136
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 10 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 3 | 8 | 11
  Black or African American | 67 | 189 | 256
  White | 355 | 693 | 1048
  More than one race | 5 | 12 | 17
  Unknown or Not Reported | 43 | 62 | 105

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Medically Attended Respiratory Syncytial Virus (RSV) Confirmed Lower Respiratory Tract Infection (LRTI)
Description: The determination of medically attended RSV LRTI is based on objective clinical LRTI criteria and RSV test results obtained from analyzing the respiratory secretions using a validated RSV real time reverse transcriptase-polymerase chain reaction (RT-PCR) assay for the detection of RSV A or RSV B subtypes. Criteria for LRTI included documented physical exam findings of rhonchi, rales, crackles, or wheeze and any of the following: increased respiratory rate at rest (for age less than (<) 2 months: greater than or equal to (>=) 60 breaths/min; 2-6 months: >= 50 breaths/min; and for > 6 months - 2 years, >= 40 breaths/min), or hypoxemia (in room air - oxygen saturation < 95% at altitudes less than or equal to (<=) 1800 meters or < 92% at altitudes > 1800 meters), or clinical signs of severe respiratory disease or dehydration secondary to inadequate oral intake due to respiratory distress (need for intravenous fluid).
Time Frame: From Day 1 through Day 151
Population: The ITT population included all participants who were randomized in the study and analyzed according to their randomized treatment group.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 50 mg
Number analyzed (Participants) | 484 | 969
Participants | 46 | 25
Statistical Analysis 1: Comparison: Placebo vs MEDI8897 50 mg; Test type: Superiority; p < 0.0001, Poisson regression; Relative Risk Reduction = 70.1, 95% CI 2-sided [52.3 to 81.2]

2. Secondary Outcome: Number of Participants Hopitalized Due to Respiratory Syncytial Virus (RSV) Confirmed Lower Respiartory Tract Infection (LRTI)
Description: A RSV hospitalization is defined as either 1) a respiratory hospitalization with a positive RSV test within 2 days of hospitalization (primary) or 2) new onset of respiratory symptoms in an already hospitalized child, with an objective measure of worsening respiratory status and positive RSV test (nosocomial).
Time Frame: From Day 1 through Day 151
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 50 mg
Number analyzed (Participants) | 484 | 969
Participants | 20 | 8
Statistical Analysis 1: Comparison: Placebo vs MEDI8897 50 mg; Test type: Superiority; p = 0.0002, Poisson regression; Relative Risk Reduction = 78.4, 95% CI 2-sided [51.9 to 90.3]

3. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) and Treatment Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are defined as events present at baseline that worsened in intensity after administration of study drug or events absent at baseline that emerged after administration of study drug.
Time Frame: From Day 1 through Day 361
Population: As-treated population included all randomized participants who received any study drug and analyzed according to the study drug they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 50 mg
Number analyzed (Participants) | 479 | 968
Participants
  TEAEs | 416 | 834
  TESAEs | 81 | 108

4. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs) and New Onset Chronic Diseases (NOCDs)
Description: An AESI was one of scientific and medical interest specific to understanding of study drug and may have required close monitoring and rapid communication by investigator to the sponsor. An AESI may be serious or non-serious. A NOCD is a newly diagnosed medical condition that is of a chronic, ongoing nature. It is observed after receiving study drug and is assessed by investigator as medically significant.
Time Frame: From Day 1 through Day 361
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 50 mg
Number analyzed (Participants) | 479 | 968
Participants
  AESIs | 3 | 5
  NOCDs | 4 | 4

5. Secondary Outcome: Serum Concentration of MEDI8897
Time Frame: Days 91, 151, and 361
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MEDI8897 50 mg
Number analyzed (Participants) | 968
mcg/mL
  Day 91: number analyzed (Participants) | 883
  Day 91 | 35.9 (10.9)
  Day 151: number analyzed (Participants) | 849
  Day 151 | 18.9 (7.4)
  Day 361: number analyzed (Participants) | 771
  Day 361 | 2.1 (1.1)

6. Secondary Outcome: Elimination Half-life (t1/2) of MEDI8897
Description: Terminal elimination half-life (t½) is the time required for half of the drug to be eliminated from the serum.
Time Frame: Day 91 through Day 361
Population: As-treated population included all randomized participants who received any study drug and analyzed according to the study drug they actually received. Participants with sufficient additional pharmacokinetics (PK) samples from unscheduled visits were analysed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | MEDI8897 50 mg
Number analyzed (Participants) | 968
Days | 59.3 (9.6)

7. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies to MEDI8897
Description: The number of participants with positive serum antibodies to MEDI8897 are reported.
Time Frame: Days 91, 151, and 361
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MEDI8897 50 mg
Number analyzed (Participants) | 479 | 968
Participants
  Day 91: number analyzed (Participants) | 455 | 890
  Day 91 | 4 | 11
  Day 151: number analyzed (Participants) | 445 | 867
  Day 151 | 6 | 17
  Day 361: number analyzed (Participants) | 418 | 847
  Day 361 | 8 | 30

ADVERSE EVENTS:
Time Frame: From Day 1 through Day 361
Description: As-treated population included all randomized participants who received any study drug and analyzed according to the study drug they actually received.
Arm/Group | Placebo | MEDI8897 50 mg
All-Cause Mortality (participants affected / at risk) | 3/479 | 2/968
Serious Adverse Events (participants affected / at risk) | 81/479 | 108/968
Other Adverse Events (participants affected / at risk) | 402/479 | 804/968
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=479) | MEDI8897 50 mg (N=968)
Anaemia neonatal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (3)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Muscular dystrophy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Deafness bilateral (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 6 (6) | 1 (1)
Malabsorption (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)
Death (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 3 (3)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 0 (0) | 1 (1)
Adenovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 21 (26) | 20 (22)
Bronchitis (Infections and infestations) | 11 (11) | 14 (16)
Croup infectious (Infections and infestations) | 0 (0) | 2 (2)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 4 (5) | 9 (9)
Gastroenteritis escherichia coli (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis adenovirus (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis rotavirus (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (2) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 13 (18) | 14 (14)
Lower respiratory tract infection viral (Infections and infestations) | 3 (5) | 5 (5)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 10 (12) | 13 (13)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia parainfluenzae viral (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 2 (2) | 2 (2)
Pneumonia viral (Infections and infestations) | 2 (2) | 7 (8)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 2 (2) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2)
Sepsis neonatal (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal scalded skin syndrome (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3)
Urinary tract infection (Infections and infestations) | 4 (5) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Palate injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Eyelid haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Infantile spasms (Nervous system disorders) | 1 (1) | 0 (0)
Intraventricular haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 2 (2)
Penile adhesion (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary vein stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=479) | MEDI8897 50 mg (N=968)
Anaemia (Blood and lymphatic system disorders) | 17 (17) | 29 (29)
Plagiocephaly (Congenital, familial and genetic disorders) | 3 (3) | 15 (15)
Abdominal pain (Gastrointestinal disorders) | 10 (10) | 5 (5)
Constipation (Gastrointestinal disorders) | 21 (24) | 34 (36)
Diarrhoea (Gastrointestinal disorders) | 49 (55) | 98 (113)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 22 (22) | 37 (38)
Teething (Gastrointestinal disorders) | 32 (35) | 62 (72)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 11 (11)
Vomiting (Gastrointestinal disorders) | 15 (17) | 40 (46)
Pyrexia (General disorders) | 63 (75) | 109 (133)
Acarodermatitis (Infections and infestations) | 8 (8) | 13 (15)
Bronchiolitis (Infections and infestations) | 42 (60) | 83 (104)
Bronchitis (Infections and infestations) | 49 (77) | 91 (150)
Candida nappy rash (Infections and infestations) | 6 (6) | 12 (14)
Conjunctivitis (Infections and infestations) | 39 (44) | 86 (94)
Croup infectious (Infections and infestations) | 6 (7) | 12 (13)
Ear infection (Infections and infestations) | 13 (21) | 23 (34)
Exanthema subitum (Infections and infestations) | 11 (11) | 21 (22)
Fungal skin infection (Infections and infestations) | 8 (8) | 5 (5)
Gastroenteritis (Infections and infestations) | 44 (49) | 115 (138)
Gastroenteritis viral (Infections and infestations) | 5 (5) | 13 (15)
Hand-foot-and-mouth disease (Infections and infestations) | 14 (14) | 36 (36)
Impetigo (Infections and infestations) | 6 (6) | 12 (12)
Laryngitis (Infections and infestations) | 10 (10) | 24 (31)
Lower respiratory tract infection (Infections and infestations) | 46 (65) | 75 (103)
Lower respiratory tract infection viral (Infections and infestations) | 6 (8) | 9 (9)
Nasopharyngitis (Infections and infestations) | 94 (158) | 164 (264)
Oral candidiasis (Infections and infestations) | 26 (26) | 36 (39)
Otitis media (Infections and infestations) | 42 (63) | 63 (87)
Otitis media acute (Infections and infestations) | 24 (33) | 51 (82)
Pharyngitis (Infections and infestations) | 27 (32) | 57 (68)
Rhinitis (Infections and infestations) | 50 (61) | 111 (145)
Tonsillitis (Infections and infestations) | 5 (6) | 16 (16)
Upper respiratory tract infection (Infections and infestations) | 169 (337) | 392 (734)
Urinary tract infection (Infections and infestations) | 7 (7) | 12 (12)
Varicella (Infections and infestations) | 11 (11) | 19 (19)
Viral rash (Infections and infestations) | 15 (16) | 32 (34)
Viral upper respiratory tract infection (Infections and infestations) | 34 (57) | 48 (75)
Arthropod bite (Injury, poisoning and procedural complications) | 6 (6) | 14 (14)
Vaccination complication (Injury, poisoning and procedural complications) | 15 (19) | 23 (28)
Irritability (Psychiatric disorders) | 7 (14) | 11 (20)
Cough (Respiratory, thoracic and mediastinal disorders) | 15 (17) | 37 (45)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 24 (27) | 71 (83)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 17 (17) | 23 (23)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 29 (34) | 63 (75)
Dermatitis (Skin and subcutaneous tissue disorders) | 15 (15) | 20 (26)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 8 (9) | 30 (34)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 36 (44) | 76 (94)
Eczema (Skin and subcutaneous tissue disorders) | 15 (15) | 34 (34)
Rash (Skin and subcutaneous tissue disorders) | 17 (18) | 43 (49)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 7 (8) | 17 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (2):
  • Study Protocol (2018-01-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT02878330/Prot_000.pdf
  • Statistical Analysis Plan (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT02878330/SAP_001.pdf